CLINICAL TRIAL: NCT01624467
Title: A Study to Determine Whether Necitumumab (IMC-11F8) Monotherapy Affects the Corrected QT (QTc) Interval in Patients With Advanced Solid Tumors
Brief Title: A Study of Necitumumab Monotherapy and the QT/QTc Interval in Patient With Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14472; CP11-1114 (Other: ImClone Systems); I4X-IE-JFCI (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-24; First posted 2012-06-20 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Solid Tumors
Keywords: Advanced Solid Tumors
MeSH Terms: interventions — necitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Necitumumab (Experimental): 800 mg necitumumab, administered once per week as an intravenous infusion (IV)
  Interventions: Biological: Necitumumab

INTERVENTIONS:
Biological: Necitumumab — 800 mg necitumumab, administered once per week IV
  Other Names: IMC-11F8; LY3012211

SUMMARY:
The purpose of this study is to determine whether treatment with necitumumab monotherapy affects the QT/QTc interval among participants with advanced solid tumors refractory to standard treatment or for which no standard treatment is available.

ELIGIBILITY:
Inclusion Criteria:

* Have documented advanced or metastatic malignant solid tumors (except for colorectal tumors with KRAS mutation) that have not responded to standard therapy or for which no standard therapy is available
* May have measurable or non-measurable disease
* Have resolution to Grade 0 or 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE 4.0) of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy
* Have an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1
* Have adequate hepatic, renal and hematologic function
* Have potassium, magnesium, and calcium within normal limits
* Subjects, if female, are surgically sterile, postmenopausal, or compliant with a highly effective contraceptive method during and for 6 months after the treatment period. If male, participants are surgically sterile or compliant with a highly effective contraceptive regimen during and for 6 months after the treatment period
* Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization

Exclusion Criteria:

* Are currently enrolled in, or discontinued a clinical trial involving an anticancer investigational product, or concurrently enrolled in any other type of medical research
* Had therapeutic radiotherapy within 14 days prior to the first dose of study therapy
* Have received necitumumab or any other monoclonal antibody (mAb) targeting the EGFR (epidermal growth factor receptor) as the most recent prior treatment
* Have documented and/or symptomatic brain or leptomeningeal metastases
* Have a clinically relevant abnormality on the ECG, preventing an accurate measurement of the QT interval
* Have current clinically-relevant coronary artery disease or uncontrolled congestive heart failure
* Have medically uncontrolled angina pectoris, or has experienced myocardial infarction within 6 months prior to the first dose of study therapy
* Have an implantable pacemaker or automatic implantable cardioverter defibrillator
* Have received sotalol within 10 days prior to the first dose of study therapy
* Have a history of risk factors for ventricular tachycardia or Torsades de pointes, history of fainting, unexplained loss of consciousness, or convulsions
* Have a history of heart failure, congestive heart failure, myocardial infarction, cardiomyopathy, hypokalemia, hypoglycemia, or hypomagnesia
* Have any evidence of conduction abnormality (eg, increased QRS complex)
* Have congenital long QT syndrome
* Have a prolonged QTc interval mean on pretreatment ECG
* Have a heart rate < 50 bpm or > 100 bpm at rest
* Are using a medication that is known to prolong the ECG QT interval, or have received a medication known to prolong the ECG QT interval within 14 days prior to first dose of study therapy
* Have a known allergy / history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of necitumumab, or a known history of severe (Grade 3-4) hypersensitivity reaction to any monoclonal antibody
* Have an ongoing or active infection (requiring treatment), including active tuberculosis or known infection with the human immunodeficiency virus
* If female, are pregnant or breastfeeding
* Have a history of significant neurological or psychiatric disorders, including dementia, seizures, or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Brunswick, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntersville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are defined as the QTc complete participants who received full doses of necitumumab for ≥1 full 6-week cycle or did not complete the first cycle because of QTc prolongation, and had pretreatment and post-infusion triplicate ECGs at the times specified in all versions of the protocol.
Groups:
- Necitumumab: 800 milligram (mg) necitumumab, administered once per week as an intravenous infusion (IV)
Period: Overall Study
Arm/Group | Necitumumab
Started | 75
Received at Least One Dose of Study Drug | 75
Completed | 44
Not Completed | 31
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 7
Not completed — Progressive Disease | 19
Not completed — Per Sponsor Requirement | 1
Not completed — Subject Withdrew from Treatment | 1

BASELINE CHARACTERISTICS:
Population: All QTc evaluable participants who received at least 1 dose of study drug.
Arm/Group | Necitumumab
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 63
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Time-Matched Baseline in QT Interval Corrected for Heart Rate (QTc)
Description: The corrected QT interval was calculated using Fridericia's correction (QTcF) from electrocardiogram (ECG) data. Each participant had triplicate QT intervals measured at each timepoint and the average was calculated for each participant at each timepoint. For each timepoint, a participant's corresponding baseline (Day -1, pretreatment) QTcF interval was subtracted from the average QTcF intervals to create the change from time-matched baseline in the QTcF interval
Time Frame: Baseline, Cycle1 Day 1, 8,15, 22, 29, and 36: Pre-infusion, End of Infusion, 1 Hour (hr), 2, 4, 24, 48, 72 hr Post Infusion
Population: QTC evaluable population: all participants who received at least 1 dose of study drug and at least 1 post-infusion ECG.
Measure: Mean (90% Confidence Interval); unit: milliseconds (msec)
Arm/Group | Necitumumab
Number analyzed (Participants) | 75
milliseconds (msec)
  Cycle 1, Day 1(D1), Pre-Infusion (n=74) | 1.00 [-0.44 to 2.44]
  Cycle 1, D1, End of Infusion (n=75) | 1.72 [0.17 to 3.28]
  Cycle 1, D1, 1 hr Post-Infusion (n=75) | 0.63 [-1.20 to 2.36]
  Cycle 1,D1, 2 hr Post-Infusion (n=75) | -0.17 [-1.84 to 1.51]
  Cycle 1,D1, 4 hr Post-Infusion (n=75) | -2.02 [-3.81 to -0.24]
  Cycle 1,D1, 24 hr Post-Infusion (n=73) | -3.12 [-4.74 to -1.50]
  Cycle 1,D1, 48 hr Post-Infusion (n=73) | -2.67 [-4.44 to -0.91]
  Cycle 1,D1, 72 hr Post-Infusion (n=72) | -1.88 [-3.87 to 0.11]
  Cycle 1, D8, Pre-Infusion (n=72) | 5.19 [2.86 to 7.52]
  Cycle 1, D8, End of Infusion (n=71) | 8.20 [5.93 to 10.47]
  Cycle 1 D8, 1 hr Post-Infusion (n=70) | 5.34 [3.12 to 7.57]
  Cycle 1, D8, 2 hr Post-Infusion (n=71) | 4.41 [2.41 to 6.40]
  Cycle 1, D8, 4 hr Post-Infusion (n=72) | 3.42 [1.45 to 5.38]
  Cycle 1, D15, Pre-Infusion (n=63) | 4.92 [2.49 to 7.52]
  Cycle 1, D15, End of Infusion (n=63) | 6.47 [4.07 to 8.88]
  Cycle 1, D15, 1 hr Post-Infusion (n=61) | 5.07 [2.57 to 7.58]
  Cycle 1, D15, 2 hr Post-Infusion (n=62) | 4.04 [1.13 to 6.95]
  Cycle 1, D15 4 hr Post-Infusion (n=62) | 3.04 [0.44 to 5.63]
  Cycle 1, D22, Pre-Infusion (n=61) | 3.87 [1.79 to 5.96]
  Cycle 1, D22, End of Infusion (n=59) | 6.89 [4.47 to 9.31]
  Cycle 1, D22, 1 hr Post-Infusion (n=59) | 5.03 [2.56 to 7.50]
  Cycle 1, D22, 2 hr Post-Infusion (n=60) | 2.48 [0.27 to 4.69]
  Cycle 1, D22 4 hr Post-Infusion (n-60) | 1.53 [-0.66 to 3.72]
  Cycle 1, D29, Pre-Infusion (n=59) | 3.68 [1.38 to 5.98]
  Cycle 1, D29, End of Infusion (n=59) | 6.95 [4.74 to 9.16]
  Cycle 1, D29, 1 hr Post-Infusion (n=59) | 3.99 [1.54 to 6.44]
  Cycle 1, D29, 2 hr Post-Infusion (n=59) | 3.25 [1.01 to 5.48]
  Cycle 1, D29, 4 hr Post-Infusion (n=59) | 1.62 [-0.40 to 3.64]
  Cycle 1, D36, Pre-Infusion (n=53) | 4.47 [2.11 to 6.84]
  Cycle 1, D36, End of Infusion (n=49) | 5.14 [2.94 to 7.34]
  Cycle 1, D36, 1 hr Post-Infusion (n=50) | 3.59 [0.82 to 6.36]
  Cycle 1, D36, 2 hr Post-Infusion (n-50) | 2.77 [0.25 to 5.29]
  Cycle 1, D36, 4 hr Post-Infusion (n=49) | 1.15 [-1.11 to 3.40]
  Cycle 1, D36, 24 hr Post-Infusion (n=49) | -0.64 [-2.83 to 1.55]
  Cycle 1, D36, 48 hr Post-Infusion (n=50) | 0.09 [-2.75 to 2.93]
  Cycle 1, D36, 72 hr Post-Infusion (n=50) | -0.20 [-2.51 to 2.12]

2. Secondary Outcome: Change From Time-Matched Baseline ≥ 25% and Absolute Value of QRS >110 Msec (Electrocardiographic Parameters: QRS Interval)
Time Frame: Baseline, Cycle1 Day 1, 8, 15, 22, 29, 36: Pre-infusion, End of Infusion, 1 Hour (hr), 2, 4, 24, 48, 72 hr Post Infusion
Population: QTC evaluable population: all participants who received at least 1 dose of study drug and at least 1 post-infusion ECG
Measure: Number; unit: participants
Arm/Group | Necitumumab
Number analyzed (Participants) | 75
participants | 0

3. Secondary Outcome: PR Change From Time-Matched Baseline ≥25% and Absolute Value of PR > 200 Msec (Electrocardiographic Parameters: PR Interval)
Time Frame: as for outcome 2
Population: QTC evaluable population: all participants who received at least 1 dose of study drug and at least 1 post-infusion ECG.
Measure: Number; unit: percentage of participants
Arm/Group | Necitumumab
Number analyzed (Participants) | 75
percentage of participants | 0

4. Secondary Outcome: Change From Time-Matched Baseline in Heart Rate (HR) (Electrocardiographic Parameters: Heart Rate [HR])
Description: Change in HR from time-matched measures performed at baseline.
Time Frame: Baseline, Cycle1 Day 36: Pre-infusion, End of Infusion, 1 Hour (hr), 2, 4, 24, 48, 72 hr Post Infusion
Population: QTC evaluable population: all participants who received at least 1 dose of study drug and at least 1 post-infusion ECG
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Necitumumab
Number analyzed (Participants) | 75
Beats/minute
  Cycle 1, D36, Pre-Infusion (n=53)) | 0.50 (10.22)
  Cycle 1, D36, End of Infusion, (n=49) | 1.92 (12.44)
  Cycle 1, D36, 1 hr Post-Infusion (n=50) | 2.73 (12.21)
  Cycle 1, D36, 2 hr Post-Infusion (n=50) | 2.02 (11.77)
  Cycle 1, D36, 4 hr Post-Infusion (n=49) | 3.36 (8.39)
  Cycle 1, D36, 24 hr Post-Infusion (n=49) | 3.56 (10.05)
  Cycle 1, D36, 48 hr Post-Infusion, (n=50) | 5.09 (10.55)
  Cycle 1, D36, 72 hr Post-Infusion (n=50) | 4.86 (12.36)
  Cycle 1, D36, 168 hr Post-Infusion (n=11) | 10.75 (15.77)

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve of Necitumumab From Zero to Infinity (AUC[0-∞])
Time Frame: Cycle1 (Days 1 and 36): Pre-infusion, 50 minutes, 1.5, 2.5, 4.5, 24, 28, 72, and 168 hours
Population: All participants who received at least one dose of study drug and had evaluable PK parameters in Cycle 1 on Days 1 and 36.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (μg*h/ml)
Groups:
- Necitumumab: Cycle 1, Day 1; Necitumumab: Cycle 1, Day 36: 800 mg necitumumab, administered once per week IV
Arm/Group | Necitumumab: Cycle 1, Day 1 | Necitumumab: Cycle 1, Day 36
Number analyzed (Participants) | 18 | 11
microgram*hour/milliliter (μg*h/ml) | 24500 (34) | 109000 (61)

6. Secondary Outcome: Pharmacokinetics: Maximum Drug Concentration (Cmax) of Necitumumab
Time Frame: Cycle 1 (Days 1 and 36); Pre-infusion, 50 minutes, 1.5, 2.5, 4.5, 24, 28, 72, and 168 hours
Population: All participants who received at least one dose of study drug and had evaluable PK parameters in Cycle 1, Days 1 and 36.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Necitumumab: Cycle 1, Day 1 | Necitumumab: Cycle 1, Day 36
Number analyzed (Participants) | 71 | 49
microgram/milliliter (μg/mL) | 270 (27) | 470 (30)

7. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR]) (Tumor Response Rate Per Response Evaluation Criteria in Solid Tumors Version 1.1 [RECIST 1.1])
Description: ORR is confirmed best overall tumor response of CR or PR. According to RECIST v1.1,CR was defined as the disappearance of all target and non-target lesions. Percentage of participants was calculated as: (total number of participants with CR or PR from start of the treatment until disease progression or recurrence)/total number of participants treated) * 100. PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD.
Time Frame: Baseline to Measured Progressive Disease (up to 21 Months)
Population: All participants who received any study drug and had CR or PR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Necitumumab
Number analyzed (Participants) | 75
percentage of participants | 2.7 [0.3 to 9.3]

8. Secondary Outcome: Number of Participants With an Incidence of Anti-Necitumumab Antibodies
Time Frame: Baseline to Post Infusion 30 Day Follow-up
Population: All participants who received at least 1 dose of study drug and had at least 1 post-infusion blood sample.
Measure: Number; unit: participants
Arm/Group | Necitumumab
Number analyzed (Participants) | 75
participants
  Overall Antibody Positive | 9
  Overall Treatment Emergent Antibody Positive | 1

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug.
Arm/Group | Necitumumab
Serious Adverse Events (participants affected / at risk) | 33/75
Other Adverse Events (participants affected / at risk) | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab (N=75)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (6)
Asthenia (General disorders) | 1 (1)
Disease recurrence (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab (N=75)
Anaemia (Blood and lymphatic system disorders) | 29 (43)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Vision blurred (Eye disorders) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 19 (32)
Nausea (Gastrointestinal disorders) | 32 (42)
Stomatitis (Gastrointestinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 21 (25)
Asthenia (General disorders) | 6 (6)
Chills (General disorders) | 10 (11)
Fatigue (General disorders) | 28 (33)
Oedema peripheral (General disorders) | 7 (8)
Pyrexia (General disorders) | 14 (16)
Urinary tract infection (Infections and infestations) | 6 (7)
Infusion related reaction (Injury, poisoning and procedural complications) | 6 (12)
Activated partial thromboplastin time prolonged (Investigations) | 4 (9)
Alanine aminotransferase increased (Investigations) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 14 (15)
Blood alkaline phosphatase increased (Investigations) | 14 (19)
Blood bilirubin increased (Investigations) | 4 (4)
Blood creatinine increased (Investigations) | 8 (13)
Electrocardiogram qt prolonged (Investigations) | 26 (61)
International normalised ratio increased (Investigations) | 4 (5)
Lymphocyte count decreased (Investigations) | 21 (59)
Weight decreased (Investigations) | 7 (9)
Decreased appetite (Metabolism and nutrition disorders) | 21 (22)
Dehydration (Metabolism and nutrition disorders) | 5 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (44)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 (34)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 26 (55)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7)
Dizziness (Nervous system disorders) | 11 (11)
Dysgeusia (Nervous system disorders) | 5 (9)
Headache (Nervous system disorders) | 44 (55)
Neuropathy peripheral (Nervous system disorders) | 4 (6)
Anxiety (Psychiatric disorders) | 8 (10)
Insomnia (Psychiatric disorders) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 25 (32)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (20)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11)
Rash (Skin and subcutaneous tissue disorders) | 31 (48)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (8)
Skin fissures (Skin and subcutaneous tissue disorders) | 6 (7)
Flushing (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days